CLINICAL TRIAL: NCT00567957
Title: Remifentanil for c-Section With General Anesthesia in Severe Preeclamptic Patients
Brief Title: Remifentanil for General Anesthesia in Preeclamptics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Tulay Ozkan Seyhan, Istanbul University- Istanbul Faculty of Medicine, Dept. of Anesthesiology
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: RP01; BYP-1833
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Pre-Eclampsia; Hypertension, Pregnancy-Induced; Pregnancy Complications
Keywords: pre-eclampsia; remifentanil; anesthesia, general; analgesics, opioid; anesthetics, intravenous; Cesarean section; newborn; maternal haemodynamic
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced; Pregnancy Complications | interventions — Remifentanil; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- C (Placebo Comparator): Saline starting before induction till entry to abdominal cavity
  Interventions: Drug: Saline
- R (Active Comparator): Remifentanil starting before induction till entry to abdominal cavity
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — 1 microg/kg iv bolus before induction followed by 0.5 microg/kg/min infusion
  Other Names: Ultiva
  Arms: R
Drug: Saline — same volume iv bolus before induction followed by same volume infusion
  Other Names: % 0.9 NaCl
  Arms: C

SUMMARY:
The purpose of this study is to determine whether remifentanil use in preeclamptic patients may blunt hemodynamic response to intubation during general anesthesia for cesarean section.

DETAILED DESCRIPTION:
General anesthesia for cesarean section involves rapid sequence induction with a muscle relaxant and barbiturate followed by endotracheal intubation. Although the use of opioids may blunt haemodynamic responses to endotracheal intubation, they are avoided in pregnant patients due to possible respiratory depressants effects on neonates.Preeclamptic patients response with exaggerated sympathoadrenal reflex to anesthesia induction and intubation. The resulting hypertension and tachycardia may result in cerebrovascular accident, pulmonary edema, arrhythmias, increased myocardial oxygen consumption and fetal hypoxia by uterine vasoconstriction. Several drugs have been used to blunt the hemodynamic disturbances to intubation, but none of them have been implicated for routine use for general anesthesia in preeclamptic patients.

Recently remifentanil has started to be used in general anesthesia of high risk obstetric patients. Remifentanil is a μ-opioid receptor agonist that is metabolized by nonspecific blood and tissue esterase hydrolysis. It has a low distribution volume with a context sensitive half life of 3 minutes. Its elimination half life is 12 minutes even after repeated boli. Previously remifentanil use in pregnant patients with cardiac pathology has been reported with minimal neonatal side effects. A randomized controlled study in normal parturient has shown that remifentanil is transferred through placenta and may cause mild neonatal depression that is easily managed. Umbilical artery and vein remifentanil concentrations has shown that remifentanil is quickly redistributed or metabolized in fetus. Thus, remifentanil may be an appropriate drug for induction and maintenance of general anesthesia in severe preeclamptic patients.

ELIGIBILITY:
Inclusion Criteria:

* Severe preeclamptic parturients with single fetus pregnancy with contraindication to regional anesthesia

Exclusion Criteria:

* Known allergy to study drugs
* Known fetal anomaly and /or gestation week and /or estimated to be nonviable (fetal weight <400 gr, gestational week<24 weeks)
* Known cardiac disease diagnosed prior to pregnancy
* Known drug abuse in the parturient
* Multifetal gestation
* Anticipated difficult airway management (mask ventilation and/or endotracheal intubation).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-02; Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | Induction to post-intubation period

SECONDARY OUTCOMES:
Heart rate | Induction to delivery
Amount of additional drugs and fluids if required | Induction to delivery
Evaluation of the newborn | Within 10 min following delivery

CONTACTS AND LOCATIONS:
Overall Officials: Tulay Ozkan Seyhan, Associate Prof, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine Anesthesiology Dept., Istanbul, Capa, Turkey (Türkiye)

REFERENCES:
- [Background] Ngan Kee WD, Khaw KS, Ma KC, Wong AS, Lee BB, Ng FF. Maternal and neonatal effects of remifentanil at induction of general anesthesia for cesarean delivery: a randomized, double-blind, controlled trial. Anesthesiology. 2006 Jan;104(1):14-20. doi: 10.1097/00000542-200601000-00004. PMID 16394684